CLINICAL TRIAL: NCT01156207
Title: Significance of Regional Ventriculo-arterial Coupling in Patients With Chronic Heart Failure: Effects of Endothelial Progenitor Cells and a Direct Renin Inhibitor
Brief Title: Significance of Regional Ventriculo-arterial Coupling in Patients With Chronic Heart Failure
Acronym: VACHF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: National Taiwan University Hospital, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NSC20110101; 201003020MB (Other Grant/Funding Number: NSC)
Record Dates: First submitted 2010-06-06; First posted 2010-07-02 (Estimated); Last update posted 2010-07-02 (Estimated); Status verified 2010-06

CONDITIONS: Heart Failure
Keywords: To establish the coupling between components of arterial load ( and components of LV myocardial deformations at baseline and 6 months after randomization.; To establish the role of EPCs on modulation of the components of arterial load and LV myocardial deformations and their coupling.
MeSH Terms: conditions — Heart Failure | interventions — aliskiren

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aliskiren (Experimental)
  Interventions: Drug: Aliskiren
- placebo (Placebo Comparator)
  Interventions: Drug: Aliskiren

INTERVENTIONS:
Drug: Aliskiren — 300mg Aliskiren qd for 6 month

SUMMARY:
Heart failure is a major health problem worldwide. Optimal treatment of this disabling and fatal condition may require functional characterization of the failed left ventricle (LV) and its interaction with the arterial system. Part of the physiological significance of the ventriculo-arterial coupling has been studied experimentally and clinically using the framework of the ratio of effective arterial elastance (Ea) to end-systolic elastance (Ees), with limited clinical applications.

From central ascending aorta to terminal arterioles, every segment of the arterial tree contributes to the arterial loads that interact and impact LV performance in both systole and diastole, leads to atrial and ventricular remodeling and hypertrophy, and results in the development of heart failure. On the other hand, the ventricular systole is a complex coordination of multi-directional myocardial fibers involving longitudinal contraction, circumferential shortening, radial thickening, twist, and torsion, the so-called LV deformations.

The purposes of the present study are to investigate the relationship between different components of hemodynamic load or arterial abnormalities and different components of LV myocardial deformations or regional LV function, the modulating effects of endothelial progenitor cells (EPCs) on the ventriculo-arterial coupling, and the therapeutic effects of aliskiren on the components of hemodynamic load and LV myocardial deformations and their couplings. The investigators will also investigate whether the ventriculo-arterial coupling, EPCs, and add-on therapy of aliskiren predict cardiovascular outcomes.

DETAILED DESCRIPTION:
In the proposed 3-year project, we hypothesize that the different components of arterial load are coupled with different components of LV function. The regional ventriculo-arterial couplings may be important in the pathogenesis of heart failure and ventricular remodeling, and in the prediction of future cardiovascular events. Therapies targeting these may play a role in the prevention and treatment of heart failure. Therefore, we will study at least 120 patients with chronic heart failure (NYHA Class II-IV) who will randomly receive a direct renin inhibitor, aliskiren, or a placebo for 6 months on top of standard therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients ≥ 18 years of age, male or female. Female patients must be either post-menopausal for one year, surgically sterile, or using effective contraceptive methods such as oral contraceptives, barrier method with spermicide or an intrauterine device.
2. Patients with a diagnosis of chronic heart failure (NYHA Class II-IV) and reduced systolic function: LVEF ≤ 45% at Visit 1 (local measurement, measured within the past 6 months assessed by echocardiogram, MUGA, CT scan, MRI or ventricular angiography).
3. NT-pro BNP ≥ 600pg/ml (BNP ≥ 150 pg/ml) at Visit 1 or NT-pro BNP ≥ 450 pg/mL (BNP (≥ 100 pg/ml) and a hospitalization for HF within last 12 months
4. Patients must be on a stable dose of either an ACE inhibitor or an ARB for at least 4 weeks prior to Visit 1.
5. Patients must be treated with a beta blocker, unless contraindicated or not tolerated, at a stable dose for at least 4 weeks prior to Visit 1.
6. Patients with documented sinus rhythm at Visit 1. -

Exclusion Criteria:

1. History of hypersensitivity to any of the study drugs.
2. Patients who require treatment with both ACEI and ARB.
3. Current acute decompensated HF (exacerbation of chronic HF manifested by signs & symptoms that may require IV therapy).
4. Symptomatic hypotension and/or less than 100 mmHg at the time of screening or less than 90 mmHg at the time of randomization.
5. eGFR < 30 ml/min/1.73m2 as measured by the MDRD formula at Visit 1 (screening) , or a > 25% decrease after 14 days of active run-in period.
6. Serum potassium > 5.0 mmol/L at screening (Visit 1).
7. Acute coronary syndrome, stroke, transient ischemic attack, cardiac, carotid or major vascular surgery, percutaneous coronary intervention (PCI) or carotid angioplasty, within the past 3 months prior to visit 1.
8. Coronary or carotid artery disease likely to require surgical or percutaneous intervention within the 6 months after Visit 1.
9. Patients with active or unstable bronchospasm or asthma (patients must be on stable regimen of respiratory medications for 1 month prior to Visit 1).
10. Right heart failure due to severe pulmonary disease.
11. Diagnosis of peripartum or chemotherapy induced cardiomyopathy within the 12 months prior to visit 1.
12. Patients with a history of heart transplant or who are on a transplant list or with left ventricular assistance device (LVAD device).
13. Documented ventricular arrhythmia with syncopal episodes within past 3 months, prior to visit 1, that is untreated.
14. Symptomatic bradycardia or second or third degree heart block without a pacemaker.
15. Implantation of a CRT (cardiac resynchronization therapy) device within the prior 3 months from visit 1 or intent to implant a CRT device.
16. Presence of hemodynamically significant mitral and/or aortic valve disease, except mitral regurgitation secondary to left ventricular dilatation.
17. Presence of other hemodynamically significant obstructive lesions of left ventricular outflow tract, including aortic and sub-aortic stenosis.
18. Severe primary pulmonary, renal or hepatic disease.
19. Presence of any other disease with a life expectancy of < 1 year.
20. Chronic long-term requirement for NSAIDs (high dose) or COX2 inhibitors, with the exception of aspirin at doses used for CV prophylaxis (≤325 mg o.d.).
21. Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of study drugs
22. Subjects get pregnant or will be pregnant within 6 months.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2010-07; Primary Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
LV systolic function, the global longitudinal strain | 1 year
  During 1-year treatment, ventricular systolic functions would be measured by using speckle tracking and presented as global longitudinal, circumferential, and radial strain at baseline and at the end of study. The changes of strain would be compared between 2 study groups.

SECONDARY OUTCOMES:
plasma NT-proBNP level | 1 year
  After 1 year, plasma NT-proBNP will be re-checked. The differences between on-treatment and baseline NT-proBNP levels will be compared between 2 groups.

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei